CLINICAL TRIAL: NCT03367403
Title: Assessment of Safety, Tolerability and Efficacy of LY3002813 in Early Symptomatic Alzheimer's Disease
Brief Title: A Study of LY3002813 in Participants With Early Symptomatic Alzheimer's Disease (TRAILBLAZER-ALZ)
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Eli Lilly and Company (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: 16933; I5T-MC-AACG (Other: Eli Lilly and Company)
Record Dates: First submitted 2017-12-05; First posted 2017-12-08 (Actual); Results first posted 2022-02-15 (Actual); Last update posted 2022-10-13 (Actual); Status verified 2022-09

CONDITIONS: Alzheimer Disease
Keywords: TRAILBLAZER-ALZ
MeSH Terms: conditions — Alzheimer Disease | interventions — donanemab; LY3202626

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (3):
- Donanemab Monotherapy (Donanemab-M) (Experimental): Participants received 700 milligram (mg) donanemab intravenously (IV) every 4 weeks (Q4W) x 3 doses, then 1400 mg donanemab IV Q4W for up to 72 weeks.
  Interventions: Drug: Donanemab
- Placebo (Placebo Comparator): Participants received placebo IV Q4W for up to 72 weeks.
  Interventions: Drug: Placebo
- Donanemab in Combination With LY3202626 (Donanemab-C) (Experimental): Participants received 700 mg donanemab IV Q4W x 3 doses, then 1400 mg donanemab IV Q4W in combination with 12 mg of LY3202626 orally for up to 72 weeks.
  As per protocol amendment (d) approved on Oct 9, 2018, donanemab in combination with LY3202626 (donanemab-C) arm discontinued as there was a low probability of identifying a statistically significant effect of 12mg of LY3202626 slowing cognitive decline.
  Interventions: Drug: Donanemab; Drug: LY3202626

INTERVENTIONS:
Drug: Donanemab — Administered IV
  Other Names: LY3002813
  Arms: Donanemab Monotherapy (Donanemab-M); Donanemab in Combination With LY3202626 (Donanemab-C)
Drug: Placebo — Administered IV
  Arms: Placebo
Drug: LY3202626 — Administered orally
  Arms: Donanemab in Combination With LY3202626 (Donanemab-C)

SUMMARY:
The purpose of this study is to evaluate the safety, tolerability and efficacy of LY3002813 in early symptomatic Alzheimer's disease.

ELIGIBILITY:
Inclusion Criteria:

* Gradual and progressive change in memory function reported by participants or informants for ≥ 6 months.
* MMSE score of 20 to 28 (inclusive) at baseline or an acceptable historical flortaucipir PET scan within 6 months prior to baseline that meets the central read criteria.
* Meet 18F flortaucipir PET scan eligibility criteria.
* Meet 18F florbetapir PET scan (central read) eligibility criteria.

Exclusion Criteria:

* Have a history of long QT syndrome.
* Have received treatment with a stable dose of an acetylcholinesterase inhibitor (AChEI) and/or memantine for less than 2 months before randomization.
* Contraindication to MRI.

Ages: 60 Years to 85 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 272 (Actual)
Dates: Start 2017-12-18 (Actual); Primary Completion 2020-12-04 (Actual); Study Completion 2021-09-21 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Call 1-877-CTLILLY (1-877-285-4559) or 1-317-615-4559 Mon - Fri 9 AM - 5 PM Eastern time (UTC/GMT - 5 hours, EST), Study Director — Eli Lilly and Company
Locations (61):
- United States (56):
  - Banner Alzheimer's Institute, Phoenix, Arizona
  - Banner Sun Health Research Institute, Sun City, Arizona
  - Neurology Center of North Orange County, Fullerton, California
  - Irvine Clinical Research Center, Irvine, California
  - Institute for Memory Impairment & Neurological Disorders, Irvine, California
  - Pharmacology Research Institute, Newport Beach, California
  - Pacific Research Network Inc, San Diego, California
  - Sharp Mesa Vista Hospital, San Diego, California
  - Syrentis Clinical Research, Santa Ana, California
  - Associated Neurologists, PC - Danbury, Danbury, Connecticut
  - KI Health Partners, LLC d/b/a NE Inst. for Clin. Res., Stamford, Connecticut
  - JEM Research Institute, Atlantis, Florida
  - Bradenton Research Center, Bradenton, Florida
  - Brain Matters Research, Delray Beach, Florida
  - Infinity Clinical Research, LLC, Hollywood, Florida
  - Jacksonville Center for Clinical Research, Jacksonville, Florida
  - Merritt Island Medical Research LLC, Merritt Island, Florida
  - Pharmax Research Clinic, Miami, Florida
  - Miami Jewish Health Systems, Miami, Florida
  - Suncoast Clinical Research, New Port Richey, Florida
  - Compass Research, Orlando, Florida
  - Palm Beach Neurological Group, Palm Beach Gardens, Florida
  - Quantum Laboratories, Pompano Beach, Florida
  - Progressive Medical Research, Port Orange, Florida
  - Intercoastal Medical Group, Sarasota, Florida
  - Axiom Research, Tampa, Florida
  - Stedman Clinical Trials, Tampa, Florida
  - Compass Research, The Villages, Florida
  - Great Lakes Clinical Trials, Chicago, Illinois
  - Alexian Brothers Medical Center, Elk Grove Village, Illinois
  - Indiana University School of Medicine, Indianapolis, Indiana
  - Josephson Wallack Munshower Neurology, Indianapolis, Indiana
  - University of Kansas Hospital, Fairway, Kansas
  - Cotton O'Neil Clinic, Topeka, Kansas
  - McLean Hospital, Belmont, Massachusetts
  - ActivMed Practices & Research, Inc, Methuen, Massachusetts
  - Boston Center for Memory, Newton, Massachusetts
  - Donald S Marks, Plymouth, Massachusetts
  - Washington University, St Louis, Missouri
  - Las Vegas Medical Research, Las Vegas, Nevada
  - Advanced Memory Research Institute of New Jersey, Toms River, New Jersey
  - Behavioral Health Center Research, Charlotte, North Carolina
  - Guilford Neurologic Associates, Greensboro, North Carolina
  - Raleigh Neurology Associates, Raleigh, North Carolina
  - Piedmont Medical Research, Winston-Salem, North Carolina
  - Insight Clinical Trials, Beachwood, Ohio
  - Ohio State University Medical Center, Columbus, Ohio
  - Neurology Diagnostics, Inc., Dayton, Ohio
  - Abington Neurological Associates, Willow Grove, Pennsylvania
  - Rhode Island Hospital, Providence, Rhode Island
  - Butler Hospital, Providence, Rhode Island
  - Texas Neurology, PA, Dallas, Texas
  - Houston Methodist, Houston, Texas
  - The Memory Clinic, Bennington, Vermont
  - Cognition Health, Fairfax, Virginia
  - National Clinical Research - Richmond, Richmond, Virginia
- Canada (5):
  - Bruyere Research Institute, Ottawa, Ontario
  - Kawartha Regional Memory Clinic, Peterborough, Ontario
  - Toronto Memory Program, Toronto, Ontario
  - Clinique de la Memoire de l'Outaouais, Gatineau, Quebec
  - DIEX Recherche Sherbrooke, Inc, Sherbrooke, Quebec

IPD SHARING:
Plan to Share IPD: Yes
Lilly provides access to the individual patient data from studies on approved medicines and indications as defined by the sponsor specific information on ClinicalStudyDataRequest.com.
  This access is provided in a timely fashion after the primary publication is accepted. Researchers need to have an approved research proposal submitted through ClinicalStudyDataRequest.com. Access to the data will be provided in a secure data sharing environment after signing a data sharing agreement.

REFERENCES:
- [Derived] Chandler JM, Lansdall CJ, Ye W, McDougall F, Belger M, Toth B, Mi X, Sink KM, Atkins AS. The Alzheimer's Disease Cooperative Study - Activities of Daily Living dependence score: revision and validation of an algorithm evaluating patient dependence across the spectrum of AD severity. J Prev Alzheimers Dis. 2025 Sep;12(8):100261. doi: 10.1016/j.tjpad.2025.100261. Epub 2025 Jul 1. PMID 40603145
- [Derived] Zimmer JA, Ardayfio P, Wang H, Khanna R, Evans CD, Lu M, Sparks J, Andersen S, Lauzon S, Nery ESM, Battioui C, Engle SE, Biffi A, Svaldi D, Salloway S, Greenberg SM, Sperling RA, Mintun M, Brooks DA, Sims JR. Amyloid-Related Imaging Abnormalities With Donanemab in Early Symptomatic Alzheimer Disease: Secondary Analysis of the TRAILBLAZER-ALZ and ALZ 2 Randomized Clinical Trials. JAMA Neurol. 2025 May 1;82(5):461-469. doi: 10.1001/jamaneurol.2025.0065. PMID 40063015
- [Derived] Klein EG, Schroeder K, Wessels AM, Phipps A, Japha M, Schilling T, Zimmer JA. How donanemab data address the coverage with evidence development questions. Alzheimers Dement. 2024 Apr;20(4):3127-3140. doi: 10.1002/alz.13700. Epub 2024 Feb 7. PMID 38323738
- [Derived] Pontecorvo MJ, Lu M, Burnham SC, Schade AE, Dage JL, Shcherbinin S, Collins EC, Sims JR, Mintun MA. Association of Donanemab Treatment With Exploratory Plasma Biomarkers in Early Symptomatic Alzheimer Disease: A Secondary Analysis of the TRAILBLAZER-ALZ Randomized Clinical Trial. JAMA Neurol. 2022 Dec 1;79(12):1250-1259. doi: 10.1001/jamaneurol.2022.3392. PMID 36251300
- [Derived] Shcherbinin S, Evans CD, Lu M, Andersen SW, Pontecorvo MJ, Willis BA, Gueorguieva I, Hauck PM, Brooks DA, Mintun MA, Sims JR. Association of Amyloid Reduction After Donanemab Treatment With Tau Pathology and Clinical Outcomes: The TRAILBLAZER-ALZ Randomized Clinical Trial. JAMA Neurol. 2022 Oct 1;79(10):1015-1024. doi: 10.1001/jamaneurol.2022.2793. PMID 36094645
- [Derived] Mintun MA, Lo AC, Duggan Evans C, Wessels AM, Ardayfio PA, Andersen SW, Shcherbinin S, Sparks J, Sims JR, Brys M, Apostolova LG, Salloway SP, Skovronsky DM. Donanemab in Early Alzheimer's Disease. N Engl J Med. 2021 May 6;384(18):1691-1704. doi: 10.1056/NEJMoa2100708. Epub 2021 Mar 13. PMID 33720637
- See also: A Study of LY3002813 in Participants With Early Symptomatic Alzheimer's Disease — https://trials.lillytrialguide.com/en-US/trial/4iGquIFHpuwam80Imyiukq

RESULTS

PARTICIPANT FLOW:
Recruitment Details: As per protocol amendment (d) approved on Oct 9, 2018, donanemab in combination with LY3202626 (donanemab-C) arm discontinued as there was a low probability of identifying a statistically significant effect of 12 milligram (mg) of LY3202626 slowing cognitive decline. Clinical efficacy was not reported for this group.
Groups:
- Donanemab Monotherapy (Donanemab-M): Participants received 700 mg donanemab intravenously (IV) every 4 weeks (Q4W) x 3 doses, then 1400 mg donanemab IV Q4W for up to 72 weeks.
- Donanemab in Combination With LY3202626 (Donanemab-C): Participants received 700 mg donanemab IV Q4W x 3 doses, then 1400 mg donanemab IV Q4W in combination with 12 mg of LY3202626 daily orally for up to 72 weeks.
Period: Overall Study
Arm/Group | Donanemab Monotherapy (Donanemab-M) | Placebo | Donanemab in Combination With LY3202626 (Donanemab-C)
Started | 131 | 126 | 15
Received at Least One Dose of Study Drug | 131 | 125 | 15
Completed | 94 | 93 | 12
Not Completed | 37 | 33 | 3
Not completed — Adverse Event | 20 | 6 | 2
Not completed — Withdrawal by Subject | 12 | 13 | 1
Not completed — Death | 1 | 2 | 0
Not completed — Physician Decision | 0 | 1 | 0
Not completed — Protocol Violation | 1 | 1 | 0
Not completed — Withdrawal Due to Caregiver Circumstances | 0 | 2 | 0
Not completed — COVID-19 | 3 | 6 | 0
Not completed — Abuse of Alcohol Intake | 0 | 1 | 0
Not completed — Subject and Study Partner do not believe study has been Beneficial and Cognition has Declined | 0 | 1 | 0

BASELINE CHARACTERISTICS:
Population: All randomized participants.
Groups:
- Donanemab Monotherapy (Donanemab-M): Participants received 700 mg donanemab IV Q4W x 3 doses, then 1400 mg donanemab IV Q4W for up to 72 weeks.
- Total: Total of all reporting groups
Arm/Group | Donanemab Monotherapy (Donanemab-M) | Placebo | Donanemab in Combination With LY3202626 (Donanemab-C) | Total
Number analyzed (Participants) | 131 | 126 | 15 | 272
Age, Continuous [Mean (Standard Deviation); unit: years] | 74.95 (5.58) | 75.35 (5.43) | 75.20 (5.99) | 75.15 (5.52)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 68 | 65 | 12 | 145
  Male | 63 | 61 | 3 | 127
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 5 | 3 | 1 | 9
  Not Hispanic or Latino | 126 | 123 | 14 | 263
  Unknown or Not Reported | 0 | 0 | 0 | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 2 | 0 | 0 | 2
  Asian | 1 | 2 | 0 | 3
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0 | 0
  Black or African American | 5 | 3 | 0 | 8
  White | 122 | 121 | 15 | 258
  More than one race | 1 | 0 | 0 | 1
  Unknown or Not Reported | 0 | 0 | 0 | 0
Region of Enrollment [Count of Participants; unit: Participants]
  Canada | 10 | 11 | 0 | 21
  United States | 121 | 115 | 15 | 251
Integrated Alzheimer's Disease Rating Scale (iADRS) [Mean (Standard Deviation); unit: score on a scale] — Integrated Alzheimer's Disease Rating Scale is used to assess whether donanemab slows down the cognitive and functional decline associated with AD compared with placebo. iADRS is a simple linear combination of 13-item alzheimer's disease assessment scale-cognitive subscale (ADAS-Cog13) and the Alzheimer's disease cooperative study-instrumental activities of daily living scale (ADCS-iADL). The scale ranges from 0 to 144, where lower scores indicate worse performance and higher score indicates better performance. Population: All randomized participants with non-missing iADRS data.
  score on a scale
    number analyzed (Participants) | 130 | 126 | 15 | 271
    (all) | 106.20 (13.03) | 105.88 (13.22) | 108.93 (10.17) | 106.20 (12.96)

OUTCOME MEASURES:

1. Primary Outcome: Change From Baseline in the Integrated Alzheimer's Disease Rating Scale (iADRS) Score
Description: Integrated Alzheimer's Disease Rating Scale is used to assess whether donanemab slows down the cognitive and functional decline associated with AD compared with placebo. iADRS is a simple linear combination of 13-item alzheimer's disease assessment scale-cognitive subscale (ADAS-Cog13) and the Alzheimer's disease cooperative study-instrumental activities of daily living scale (ADCS-iADL). The scale ranges from 0 to 144, where lower scores indicate worse performance and higher score indicates better performance. Least Squares (LS) Mean value was controlled for fixed, categorical effects of treatment, visit and treatment-by-visit interaction, pooled investigator, acetylcholinesterase inhibitor (AChEI) and/or memantine use at baseline, as well as the continuous, fixed covariates of baseline, baseline-by-visit, and age at baseline.
Time Frame: Baseline, 76 Weeks
Population: All participants randomized to donanemab monotherapy or placebo with a baseline and at least one non-missing postbaseline iADRS data. Per protocol, outcomes were analyzed by comparing donanemab Monotherapy (Donanemab-M) and placebo.
Measure: Least Squares Mean (Standard Error); unit: score on a scale
Arm/Group | Donanemab Monotherapy (Donanemab-M) | Placebo
Number analyzed (Participants) | 93 | 91
score on a scale | -6.86 (1.135) | -10.06 (1.141)
Statistical Analysis 1: Comparison: Donanemab Monotherapy (Donanemab-M) vs Placebo; Test type: Superiority; p = 0.042, Mixed Models Analysis; Mean Difference (Final Values) = 3.20, 95% CI 2-sided [0.12 to 6.27], Standard Error of Mean 1.560

2. Secondary Outcome: Change From Baseline in the 13-item Alzheimer's Disease Assessment Scale-Cognitive Subscale (ADAS-Cog13) Score
Description: The ADAS is a rater administered instrument that was designed to assess the severity of the dysfunction in the cognitive and noncognitive behaviors characteristic of persons with AD. The cognitive subscale of the ADAS consists of 13 items assessing areas of cognitive function most typically impaired in AD: orientation, verbal memory, language, praxis, delayed free recall, digit cancellation. The ADAS--Cog13 scale ranges from 0 to 85. Higher scores indicate greater disease severity. LS Mean value was controlled for fixed, categorical effects of treatment, visit and treatment-by-visit interaction, pooled investigator, AChEI and/or memantine use at baseline, as well as the continuous, fixed covariates of baseline, baseline-by-visit, and age at baseline.
Time Frame: Baseline, 76 Weeks
Population: All randomized participants who received at least one dose of study drug with baseline and post-baseline ADAS-Cog13 data. Per protocol, outcomes were analyzed by comparing donanemab Monotherapy (Donanemab-M) and placebo.
Measure: Least Squares Mean (Standard Error); unit: score on a scale
Arm/Group | Donanemab Monotherapy (Donanemab-M) | Placebo
Number analyzed (Participants) | 93 | 93
score on a scale | 2.91 (0.659) | 4.77 (0.660)
Statistical Analysis 1: Comparison: Donanemab Monotherapy (Donanemab-M) vs Placebo; Test type: Superiority; p = 0.040, Mixed Models Analysis; Mean Difference (Final Values) = -1.86, 95% CI 2-sided [-3.63 to -0.09], Standard Error of Mean 0.898

3. Secondary Outcome: Change From Baseline in the Clinical Dementia Rating Scale Sum of Boxes (CDR-SB) Score
Description: CDR-SB is a semi-structured interview of participants and their caregivers. Participant's cognitive status is rated across 6 domains of functioning, including memory, orientation, judgment/problem solving, community affairs, home/hobbies, and personal care. Severity score assigned for each of 6 domains; Total score (SB) ranges from 0 to 18. Higher scores indicate greater disease severity. LS Mean value was controlled for fixed, categorical effects of treatment, visit and treatment-by-visit interaction, pooled investigator, AChEI and/or memantine use at baseline, as well as the continuous, fixed covariates of baseline, baseline-by-visit, and age at baseline.
Time Frame: Baseline, 76 Weeks
Population: All randomized participants who received at least one dose of study drug with baseline and post-baseline CDR-SB data. Per protocol, outcomes were analyzed by comparing donanemab Monotherapy (Donanemab-M) and placebo.
Measure: Least Squares Mean (Standard Error); unit: score on a scale
Arm/Group | Donanemab Monotherapy (Donanemab-M) | Placebo
Number analyzed (Participants) | 93 | 90
score on a scale | 1.22 (0.176) | 1.58 (0.178)
Statistical Analysis 1: Comparison: Donanemab Monotherapy (Donanemab-M) vs Placebo; Test type: Superiority; p = 0.139, Mixed Models Analysis; Mean Difference (Final Values) = -0.36, 95% CI 2-sided [-0.83 to 0.12], Standard Error of Mean 0.239

4. Secondary Outcome: Change From Baseline in the Mini Mental State Examination (MMSE) Score
Description: MMSE is a brief screening instrument used to assess cognitive function (orientation, memory, attention, ability to name objects, follow verbal/written commands, write a sentence, and copy figures). Total score ranges from 0 to 30; lower score indicates greater disease severity. LS Mean value was controlled for fixed, categorical effects of treatment, visit and treatment-by-visit interaction, pooled investigator, AChEI and/or memantine use at baseline, as well as the continuous, fixed covariates of baseline, baseline-by-visit, and age at baseline.
Time Frame: Baseline, 76 Weeks
Population: All randomized participants who received at least one dose of study drug with baseline and post-baseline MMSE data. Per protocol, outcomes were analyzed by comparing donanemab Monotherapy (Donanemab-M) and placebo.
Measure: Least Squares Mean (Standard Error); unit: score on a scale
Arm/Group | Donanemab Monotherapy (Donanemab-M) | Placebo
Number analyzed (Participants) | 91 | 90
score on a scale | -2.35 (0.386) | -2.98 (0.390)
Statistical Analysis 1: Comparison: Donanemab Monotherapy (Donanemab-M) vs Placebo; Test type: Superiority; p = 0.227, Mixed Models Analysis; Mean Difference (Final Values) = 0.64, 95% CI 2-sided [-0.40 to 1.67], Standard Error of Mean 0.525

5. Secondary Outcome: Change From Baseline in Alzheimer's Disease Cooperative Study-Instrumental Activities of Daily Living Scale (ADCS-iADL) Score
Description: The ADCS-ADL is a 23-item inventory developed as a rater-administered questionnaire answered by the participant's caregiver. The ADCS-ADL measures both basic and instrumental activities (instrumental activity items 6a, 7-23) of daily living by participants. The range for the ADCS-iADL is 0-59 with higher scores reflecting better performance. LS Mean value was controlled for fixed, categorical effects of treatment, visit and treatment-by-visit interaction, pooled investigator, AChEI and/or memantine use at baseline, as well as the continuous, fixed covariates of baseline, baseline-by-visit, and age at baseline.
Time Frame: Baseline, 76 Weeks
Population: All randomized participants who received at least one dose of study drug with baseline and post-baseline ADCS-iADL data. Per protocol, outcomes were analyzed by comparing donanemab Monotherapy (Donanemab-M) and placebo.
Measure: Least Squares Mean (Standard Error); unit: score on a scale
Arm/Group | Donanemab Monotherapy (Donanemab-M) | Placebo
Number analyzed (Participants) | 93 | 91
score on a scale | -3.98 (0.738) | -5.20 (0.743)
Statistical Analysis 1: Comparison: Donanemab Monotherapy (Donanemab-M) vs Placebo; Test type: Superiority; p = 0.230, Mixed Models Analysis; Mean Difference (Final Values) = 1.21, 95% CI 2-sided [-0.77 to 3.20], Standard Error of Mean 1.009

6. Secondary Outcome: Change From Baseline in Brain Amyloid Plaque Deposition as Measured by Florbetapir F18 Positron Emission Tomography (PET) Scan
Description: Florbetapir PET imaging was used as a quantitative amyloid biomarker. Florbetapir PET scans at baseline and at 76 weeks after the first treatment were used to quantitatively estimate change in amyloid plaques. Quantitative amyloid burden was first formalized as the average Standardized Uptake Value Ratio (SUVR) in six predetermined cortical areas of the brain relative to the cerebellum as a reference region. Larger SUVR reflects the larger cortical amyloid burden relative to cerebellum. SUVR values were further calibrated to a centiloid (CL) scale. The Centiloid scale anchor points are 0 and 100, where 0 represents a high-certainty amyloid negative scan and 100 represents the amount of global amyloid deposition found in a typical AD scan. Least Squares mean change was controlled for fixed, categorical effects of treatment, visit and treatment-by-visit interaction, as well as the continuous, fixed covariates of baseline, baseline-by-visit, and age at baseline.
Time Frame: Baseline, 76 Weeks
Population: All randomized participants who received at least one dose of study drug with baseline and post-baseline PET amyloid data. Per protocol, outcomes were analyzed by comparing donanemab Monotherapy (Donanemab-M) and placebo.
Measure: Least Squares Mean (Standard Error); unit: centiloids
Arm/Group | Donanemab Monotherapy (Donanemab-M) | Placebo
Number analyzed (Participants) | 90 | 91
centiloids | -84.13 (2.723) | 0.93 (2.739)
Statistical Analysis 1: Comparison: Donanemab Monotherapy (Donanemab-M) vs Placebo; Test type: Superiority; p < 0.001, Mixed Models Analysis; Mean Difference (Final Values) = -85.06, 95% CI 2-sided [-92.68 to -77.43], Standard Error of Mean 3.867

7. Secondary Outcome: Change From Baseline in Brain Tau Deposition as Measured by Flortaucipir F18 PET Scan
Description: Flortaucipir PET imaging was used as a quantitative tau biomarker. Flortaucipir PET scans at baseline and at 76 weeks after the first treatment were used to quantitatively estimate change in aggregated tau neurofibrillary tangles (NFTs). Quantitative tau burden was formalized using two measures: weighted average Standardized Uptake Value Ratio (MUBADA SUVR) in the brain relative to the cerebellum gray as a reference region and the global tau load (TauL) generated using a TauIQ method. Larger weighted average SUVR reflects the larger cortical tau burden relative to cerebellum gray. The TauIQ method quantifies the spatiotemporal accumulation pattern of tau and larger TauL value reflects the larger global tau level in the brain as determined using a TauIQ mathematical framework. Least Squares mean change was controlled for baseline + age + treatment (Type III sum of squares).
Time Frame: Baseline, 76 Weeks
Population: All randomized participants who received at least one dose of study drug with non-missing baseline and at least one non-missing post-baseline PET tau data. Per protocol, outcomes were analyzed by comparing donanemab Monotherapy (Donanemab-M) and placebo.
Measure: Least Squares Mean (Standard Error); unit: standardized uptake value ratio (SUVR)
Arm/Group | Donanemab Monotherapy (Donanemab-M) | Placebo
Number analyzed (Participants) | 90 | 87
standardized uptake value ratio (SUVR)
  Tau-IQ | 0.55 (0.007) | 0.55 (0.007)
  MUBADA-Cerebellum: number analyzed (Participants) | 89 | 84
  MUBADA-Cerebellum | 1.54 (0.009) | 1.58 (0.010)
Statistical Analysis 1: Comparison: Donanemab Monotherapy (Donanemab-M) vs Placebo; Tau-IQ; Test type: Superiority; p = 0.560, ANCOVA; Mean Difference (Final Values) = 0.01, 95% CI 2-sided [-0.01 to 0.03]
Statistical Analysis 2: Comparison: Donanemab Monotherapy (Donanemab-M) vs Placebo; MUBADA-Cerebellum; Test type: Superiority; p = 0.012, ANCOVA; Mean Difference (Final Values) = 0.035, 95% CI 2-sided [0.007 to 0.062]

8. Secondary Outcome: Change From Baseline in Brain Volume as Measured by Volumetric Magnetic Resonance Imaging (vMRI)
Description: MRI scans at baseline and at 76 weeks after the first treatment were used to quantitatively estimate change in brain atrophy. Volumetric MRI (vMRI) parameters were measured in 14 brain regions: bilateral cortical, bilateral entorhinal cortex, bilateral hippocampus, bilateral inferior parietal lobe, bilateral isthmus cingulate, bilateral lateral parietal lobe, bilateral medial temporal lobe, bilateral precuneus, bilateral prefrontal lobe, bilateral superior temporal lobe, bilateral ventricles, bilateral whole brain, bilateral whole temporal lobe, and bilateral white matter. The atrophy was assessed by tensor-based morphometry, which captures volume changes within the deformation map. LS Mean value was controlled for fixed, categorical effects of treatment, visit and treatment-by-visit interaction, fixed covariates of baseline, and age at baseline.
Time Frame: Baseline, 76 Weeks
Population: All randomized participants who received at least one dose of study drug with non-missing baseline value and at least one non-missing post-baseline value. Per protocol, outcomes were analyzed by comparing donanemab monotherapy (Donanemab-M) and placebo.
Measure: Least Squares Mean (Standard Error); unit: cubic centimeter (cm^3)
Arm/Group | Donanemab Monotherapy (Donanemab-M) | Placebo
Number analyzed (Participants) | 82 | 83
cubic centimeter (cm^3)
  Bilateral Cortical | -11.18 (0.447) | -8.51 (0.445)
  Bilateral Entorhinal Cortex | -0.17 (0.008) | -0.17 (0.008)
  Bilateral Hippocampus | -0.22 (0.013) | -0.22 (0.013)
  Bilateral Inferior Parietal Lobe | -0.53 (0.033) | -0.45 (0.033)
  Bilateral Isthmuscingulate | -0.15 (0.008) | -0.13 (0.008)
  Bilateral Lateral Parietal Lobe | -1.60 (0.084) | -1.26 (0.083)
  Bilateral Medial Temporal Lobe | -0.73 (0.025) | -0.72 (0.025)
  Bilateral Precuneus | -0.71 (0.032) | -0.55 (0.032)
  Bilateral Prefrontal Lobe | -1.50 (0.081) | -1.11 (0.080)
  Bilateral Superior Temporal Lobe | -0.73 (0.031) | -0.52 (0.031)
  Bilateral Ventricles | 8.66 (0.412) | 6.38 (0.410)
  Bilateral Whole Brain | -24.53 (1.077) | -19.95 (1.072)
  Bilateral Whole Temporal Lobe | -3.52 (0.126) | -2.84 (0.126)
  Bilateral White Matter | -11.03 (0.700) | -8.75 (0.696)
Statistical Analysis 1: Comparison: Donanemab Monotherapy (Donanemab-M) vs Placebo; Bilateral Cortical; Test type: Superiority; p < 0.001, Mixed Models Analysis; Mean Difference (Final Values) = -2.67, 95% CI 2-sided [-3.92 to -1.43], Standard Error of Mean 0.631
Statistical Analysis 2: Comparison: Donanemab Monotherapy (Donanemab-M) vs Placebo; Bilateral Entorhinal Cortex; Test type: Superiority; p = 0.916, Mixed Models Analysis; Mean Difference (Final Values) = -0.00, 95% CI 2-sided [-0.02 to 0.02], Standard Error of Mean 0.011
Statistical Analysis 3: Comparison: Donanemab Monotherapy (Donanemab-M) vs Placebo; Test type: Superiority — Bilateral Hippocampus; p = 0.771, Mixed Models Analysis; Mean Difference (Final Values) = 0.01, 95% CI 2-sided [-0.03 to 0.04], Standard Error of Mean 0.019
Statistical Analysis 4: Comparison: Donanemab Monotherapy (Donanemab-M) vs Placebo; Bilateral Inferior Parietal Lobe; Test type: Superiority; p = 0.094, Mixed Models Analysis; Mean Difference (Final Values) = -0.08, 95% CI 2-sided [-0.17 to 0.01], Standard Error of Mean 0.047
Statistical Analysis 5: Comparison: Donanemab Monotherapy (Donanemab-M) vs Placebo; Bilateral Isthmuscingulate; Test type: Superiority; p = 0.052, Mixed Models Analysis; Mean Difference (Final Values) = -0.02, 95% CI 2-sided [-0.04 to 0.00], Standard Error of Mean 0.011
Statistical Analysis 6: Comparison: Donanemab Monotherapy (Donanemab-M) vs Placebo; Bilateral Lateral Parietal Lobe; Test type: Superiority; p = 0.005, Mixed Models Analysis; Mean Difference (Final Values) = -0.34, 95% CI 2-sided [-0.57 to -0.11], Standard Error of Mean 0.118
Statistical Analysis 7: Comparison: Donanemab Monotherapy (Donanemab-M) vs Placebo; Bilateral Medial Temporal Lobe; Test type: Superiority; p = 0.731, Mixed Models Analysis; Mean Difference (Final Values) = -0.01, 95% CI 2-sided [-0.08 to 0.06], Standard Error of Mean 0.036
Statistical Analysis 8: Comparison: Donanemab Monotherapy (Donanemab-M) vs Placebo; Bilateral Precuneus; Test type: Superiority; p < 0.001, Mixed Models Analysis; Mean Difference (Final Values) = -0.16, 95% CI 2-sided [-0.25 to -0.07], Standard Error of Mean 0.046
Statistical Analysis 9: Comparison: Donanemab Monotherapy (Donanemab-M) vs Placebo; Bilateral Prefrontal Lobe; Test type: Superiority; p < 0.001, Mixed Models Analysis; Mean Difference (Final Values) = -0.40, 95% CI 2-sided [-0.62 to -0.17], Standard Error of Mean 0.114
Statistical Analysis 10: Comparison: Donanemab Monotherapy (Donanemab-M) vs Placebo; Bilateral Superior Temporal Lobe; Test type: Superiority; p < 0.001, Mixed Models Analysis; Mean Difference (Final Values) = -0.21, 95% CI 2-sided [-0.30 to -0.12], Standard Error of Mean 0.044
Statistical Analysis 11: Comparison: Donanemab Monotherapy (Donanemab-M) vs Placebo; Bilateral Ventricles; Test type: Superiority; p < 0.001, Mixed Models Analysis; Mean Difference (Final Values) = 2.28, 95% CI 2-sided [1.14 to 3.43], Standard Error of Mean 0.581
Statistical Analysis 12: Comparison: Donanemab Monotherapy (Donanemab-M) vs Placebo; Bilateral Whole Brain; Test type: Superiority; p = 0.003, Mixed Models Analysis; Mean Difference (Final Values) = -4.58, 95% CI 2-sided [-7.58 to -1.59], Standard Error of Mean 1.519
Statistical Analysis 13: Comparison: Donanemab Monotherapy (Donanemab-M) vs Placebo; Bilateral Whole Temporal Lobe; Test type: Superiority; p < 0.001, Mixed Models Analysis; Mean Difference (Final Values) = -0.68, 95% CI 2-sided [-1.03 to -0.33], Standard Error of Mean 0.178
Statistical Analysis 14: Comparison: Donanemab Monotherapy (Donanemab-M) vs Placebo; Bilateral White Matter; Test type: Superiority; p = 0.022, Mixed Models Analysis; Mean Difference (Final Values) = -2.28, 95% CI 2-sided [-4.23 to -0.33], Standard Error of Mean 0.987

ADVERSE EVENTS:
Time Frame: Baseline Up To 124 Weeks
Description: All randomized participants who received at least one dose of study drug.
Arm/Group | Donanemab Monotherapy (Donanemab-M) | Placebo | Donanemab in Combination With LY3202626 (Donanemab-C)
All-Cause Mortality (participants affected / at risk) | 1/131 | 2/125 | 0/15
Serious Adverse Events (participants affected / at risk) | 26/131 | 25/125 | 3/15
Other Adverse Events (participants affected / at risk) | 118/131 | 112/125 | 15/15
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk, or affected / at risk where a term's number at risk differs (number of events):
Term (organ system) | Donanemab Monotherapy (Donanemab-M) (N=131) | Placebo (N=125) | Donanemab in Combination With LY3202626 (Donanemab-C) (N=15)
Anaemia (Blood and lymphatic system disorders) | 1 (2) | 0 (0) | 0 (0)
Acute myocardial infarction (Cardiac disorders) | 0 (0) | 2 (2) | 0 (0)
Atrial fibrillation (Cardiac disorders) | 1 (1) | 0 (0) | 0 (0)
Atrial flutter (Cardiac disorders) | 0 (0) | 1 (1) | 0 (0)
Atrioventricular block complete (Cardiac disorders) | 0 (0) | 1 (1) | 0 (0)
Cardiac arrest (Cardiac disorders) | 0 (0) | 1 (1) | 0 (0)
Cardiac failure chronic (Cardiac disorders) | 0 (0) | 1 (1) | 0 (0)
Sinus node dysfunction (Cardiac disorders) | 1 (1) | 0 (0) | 0 (0)
Vertigo (Ear and labyrinth disorders) | 0 (0) | 0 (0) | 1 (1)
Duodenal ulcer haemorrhage (Gastrointestinal disorders) | 1 (1) | 0 (0) | 0 (0)
Mouth swelling (Gastrointestinal disorders) | 0 (0) | 1 (1) | 0 (0)
Nausea (Gastrointestinal disorders) | 0 (0) | 0 (0) | 1 (1)
Small intestinal obstruction (Gastrointestinal disorders) | 1 (1) | 0 (0) | 0 (0)
Asthenia (General disorders) | 0 (0) | 1 (1) | 0 (0)
Death (General disorders) | 1 (1) | 0 (0) | 0 (0)
Non-cardiac chest pain (General disorders) | 0 (0) | 1 (1) | 0 (0)
Bile duct stone (Hepatobiliary disorders) | 0 (0) | 1 (1) | 0 (0)
Bacterial sepsis (Infections and infestations) | 1 (1) | 0 (0) | 0 (0)
Clostridium difficile colitis (Infections and infestations) | 1 (1) | 0 (0) | 0 (0)
Covid-19 pneumonia (Infections and infestations) | 1 (1) | 0 (0) | 0 (0)
Gastroenteritis (Infections and infestations) | 1 (1) | 0 (0) | 0 (0)
Pneumonia (Infections and infestations) | 5 (5) | 1 (1) | 0 (0)
Staphylococcal infection (Infections and infestations) | 0 (0) | 1 (1) | 0 (0)
Urinary tract infection (Infections and infestations) | 0 (0) | 1 (1) | 1 (1)
Urosepsis (Infections and infestations) | 0 (0) | 0 (0) | 1 (1)
Cervical vertebral fracture (Injury, poisoning and procedural complications) | 1 (1) | 0 (0) | 0 (0)
Extradural haematoma (Injury, poisoning and procedural complications) | 1 (1) | 0 (0) | 0 (0)
Fall (Injury, poisoning and procedural complications) | 0 (0) | 1 (1) | 0 (0)
Hip fracture (Injury, poisoning and procedural complications) | 1 (1) | 2 (2) | 0 (0)
Humerus fracture (Injury, poisoning and procedural complications) | 0 (0) | 1 (1) | 0 (0)
Infusion related reaction (Injury, poisoning and procedural complications) | 2 (2) | 0 (0) | 0 (0)
Jaw fracture (Injury, poisoning and procedural complications) | 1 (1) | 0 (0) | 0 (0)
Pelvic fracture (Injury, poisoning and procedural complications) | 0 (0) | 1 (1) | 0 (0)
Road traffic accident (Injury, poisoning and procedural complications) | 0 (0) | 1 (1) | 0 (0)
Seroma (Injury, poisoning and procedural complications) | 0 (0) | 1 (1) | 0 (0)
Subdural haematoma (Injury, poisoning and procedural complications) | 1 (1) | 0 (0) | 0 (0)
Upper limb fracture (Injury, poisoning and procedural complications) | 0 (0) | 1 (1) | 0 (0)
Dehydration (Metabolism and nutrition disorders) | 2 (2) | 1 (2) | 1 (1)
Diabetes mellitus (Metabolism and nutrition disorders) | 0 (0) | 1 (1) | 0 (0)
Gout (Metabolism and nutrition disorders) | 0 (0) | 1 (1) | 0 (0)
Type 2 diabetes mellitus (Metabolism and nutrition disorders) | 0 (0) | 0 (0) | 1 (1)
Intervertebral disc degeneration (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 1 (1)
Osteoarthritis (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1) | 0 (0)
Rheumatoid arthritis (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0) | 0 (0)
Bladder squamous cell carcinoma stage ii (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 1 (1) | 0 (0)
Breast cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0) | 0 (0)
Non-small cell lung cancer stage ii (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0) | 0 (0)
Prostate cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1/63 (1) | 0/61 (0) | 0/3 (0)
Squamous cell carcinoma of skin (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 1 (1) | 0 (0)
Amyloid related imaging abnormality-oedema/effusion (Nervous system disorders) | 2 (2) | 0 (0) | 0 (0)
Cerebrovascular accident (Nervous system disorders) | 1 (1) | 0 (0) | 0 (0)
Cognitive disorder (Nervous system disorders) | 0 (0) | 1 (1) | 0 (0)
Dizziness (Nervous system disorders) | 0 (0) | 1 (1) | 0 (0)
Encephalopathy (Nervous system disorders) | 1 (1) | 0 (0) | 0 (0)
Motor neurone disease (Nervous system disorders) | 0 (0) | 1 (1) | 0 (0)
Subarachnoid haemorrhage (Nervous system disorders) | 0 (0) | 0 (0) | 1 (1)
Syncope (Nervous system disorders) | 2 (2) | 1 (1) | 0 (0)
Agitation (Psychiatric disorders) | 0 (0) | 1 (1) | 0 (0)
Anxiety (Psychiatric disorders) | 0 (0) | 0 (0) | 1 (1)
Brief psychotic disorder without marked stressors (Psychiatric disorders) | 0 (0) | 1 (1) | 0 (0)
Confusional state (Psychiatric disorders) | 0 (0) | 1 (1) | 0 (0)
Mental disorder due to a general medical condition (Psychiatric disorders) | 0 (0) | 0 (0) | 1 (1)
Psychotic disorder (Psychiatric disorders) | 0 (0) | 1 (1) | 0 (0)
Acute kidney injury (Renal and urinary disorders) | 1 (1) | 0 (0) | 0 (0)
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 1 (1)
Pharyngeal swelling (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1) | 0 (0)
Pneumonia aspiration (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1) | 0 (0)
Pulmonary embolism (Respiratory, thoracic and mediastinal disorders) | 2 (2) | 0 (0) | 0 (0)
Drug eruption (Skin and subcutaneous tissue disorders) | 1 (1) | 0 (0) | 0 (0)
Aortic aneurysm (Vascular disorders) | 0 (0) | 1 (1) | 0 (0)
Hypertension (Vascular disorders) | 0 (0) | 1 (1) | 0 (0)
Hypotension (Vascular disorders) | 0 (0) | 1 (1) | 0 (0)
Orthostatic hypertension (Vascular disorders) | 1 (1) | 0 (0) | 0 (0)
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk, or affected / at risk where a term's number at risk differs (number of events):
Term (organ system) | Donanemab Monotherapy (Donanemab-M) (N=131) | Placebo (N=125) | Donanemab in Combination With LY3202626 (Donanemab-C) (N=15)
Anaemia (Blood and lymphatic system disorders) | 0 (0) | 2 (2) | 0 (0)
Anaemia of chronic disease (Blood and lymphatic system disorders) | 1 (1) | 0 (0) | 0 (0)
Leukopenia (Blood and lymphatic system disorders) | 0 (0) | 2 (2) | 0 (0)
Neutropenia (Blood and lymphatic system disorders) | 0 (0) | 2 (2) | 0 (0)
Thrombocytopenia (Blood and lymphatic system disorders) | 0 (0) | 2 (2) | 0 (0)
Angina pectoris (Cardiac disorders) | 0 (0) | 2 (2) | 0 (0)
Aortic valve stenosis (Cardiac disorders) | 0 (0) | 1 (1) | 0 (0)
Atrial fibrillation (Cardiac disorders) | 2 (2) | 3 (3) | 0 (0)
Atrial flutter (Cardiac disorders) | 1 (1) | 2 (2) | 0 (0)
Bradycardia (Cardiac disorders) | 2 (2) | 0 (0) | 0 (0)
Bundle branch block left (Cardiac disorders) | 1 (1) | 0 (0) | 0 (0)
Bundle branch block right (Cardiac disorders) | 1 (1) | 1 (1) | 0 (0)
Cardiac failure congestive (Cardiac disorders) | 0 (0) | 1 (3) | 0 (0)
Chronic left ventricular failure (Cardiac disorders) | 0 (0) | 1 (1) | 0 (0)
Diastolic dysfunction (Cardiac disorders) | 0 (0) | 1 (1) | 0 (0)
Mitral valve incompetence (Cardiac disorders) | 1 (1) | 0 (0) | 0 (0)
Palpitations (Cardiac disorders) | 2 (3) | 1 (1) | 0 (0)
Right ventricular enlargement (Cardiac disorders) | 0 (0) | 1 (1) | 0 (0)
Sinus arrest (Cardiac disorders) | 1 (1) | 0 (0) | 0 (0)
Sinus arrhythmia (Cardiac disorders) | 1 (1) | 0 (0) | 0 (0)
Sinus bradycardia (Cardiac disorders) | 2 (2) | 0 (0) | 0 (0)
Tachycardia (Cardiac disorders) | 1 (1) | 0 (0) | 0 (0)
Ventricular extrasystoles (Cardiac disorders) | 1 (1) | 1 (1) | 0 (0)
Arteriovenous malformation (Congenital, familial and genetic disorders) | 1 (1) | 0 (0) | 0 (0)
Cerumen impaction (Ear and labyrinth disorders) | 0 (0) | 2 (2) | 0 (0)
Hypoacusis (Ear and labyrinth disorders) | 1 (1) | 0 (0) | 0 (0)
Tinnitus (Ear and labyrinth disorders) | 2 (2) | 3 (3) | 0 (0)
Vertigo (Ear and labyrinth disorders) | 0 (0) | 2 (2) | 0 (0)
Goitre (Endocrine disorders) | 0 (0) | 1 (1) | 0 (0)
Hypothyroidism (Endocrine disorders) | 0 (0) | 2 (2) | 0 (0)
Cataract (Eye disorders) | 4 (6) | 0 (0) | 0 (0)
Conjunctival haemorrhage (Eye disorders) | 2 (2) | 0 (0) | 0 (0)
Corneal erosion (Eye disorders) | 0 (0) | 1 (1) | 0 (0)
Dry age-related macular degeneration (Eye disorders) | 1 (1) | 0 (0) | 0 (0)
Dry eye (Eye disorders) | 1 (1) | 0 (0) | 0 (0)
Eye pain (Eye disorders) | 0 (0) | 1 (1) | 0 (0)
Eye pruritus (Eye disorders) | 0 (0) | 0 (0) | 1 (1)
Eyelid ptosis (Eye disorders) | 1 (1) | 0 (0) | 0 (0)
Glaucoma (Eye disorders) | 1 (1) | 0 (0) | 0 (0)
Lacrimation increased (Eye disorders) | 1 (1) | 0 (0) | 0 (0)
Ocular hyperaemia (Eye disorders) | 1 (1) | 0 (0) | 0 (0)
Optic disc haemorrhage (Eye disorders) | 1 (1) | 0 (0) | 0 (0)
Photophobia (Eye disorders) | 1 (1) | 0 (0) | 0 (0)
Photopsia (Eye disorders) | 1 (1) | 0 (0) | 0 (0)
Retinal artery occlusion (Eye disorders) | 0 (0) | 0 (0) | 1 (1)
Retinal detachment (Eye disorders) | 0 (0) | 1 (1) | 0 (0)
Visual impairment (Eye disorders) | 1 (1) | 1 (1) | 0 (0)
Vitreous degeneration (Eye disorders) | 1 (1) | 0 (0) | 0 (0)
Abdominal discomfort (Gastrointestinal disorders) | 0 (0) | 1 (1) | 0 (0)
Abdominal pain (Gastrointestinal disorders) | 2 (2) | 0 (0) | 0 (0)
Anal incontinence (Gastrointestinal disorders) | 2 (2) | 0 (0) | 0 (0)
Ascites (Gastrointestinal disorders) | 0 (0) | 1 (1) | 0 (0)
Chapped lips (Gastrointestinal disorders) | 1 (1) | 0 (0) | 0 (0)
Colitis ischaemic (Gastrointestinal disorders) | 1 (1) | 0 (0) | 0 (0)
Constipation (Gastrointestinal disorders) | 3 (3) | 3 (3) | 1 (1)
Dental caries (Gastrointestinal disorders) | 0 (0) | 2 (2) | 0 (0)
Diarrhoea (Gastrointestinal disorders) | 11 (14) | 5 (5) | 0 (0)
Dry mouth (Gastrointestinal disorders) | 1 (1) | 0 (0) | 0 (0)
Dysphagia (Gastrointestinal disorders) | 3 (3) | 1 (1) | 0 (0)
Enterocolitis (Gastrointestinal disorders) | 0 (0) | 0 (0) | 1 (1)
Faeces soft (Gastrointestinal disorders) | 1 (1) | 0 (0) | 0 (0)
Gastrooesophageal reflux disease (Gastrointestinal disorders) | 2 (2) | 3 (3) | 0 (0)
Haematemesis (Gastrointestinal disorders) | 0 (0) | 1 (1) | 0 (0)
Haematochezia (Gastrointestinal disorders) | 0 (0) | 1 (1) | 0 (0)
Hiatus hernia (Gastrointestinal disorders) | 2 (2) | 0 (0) | 0 (0)
Large intestine polyp (Gastrointestinal disorders) | 0 (0) | 2 (2) | 1 (1)
Melaena (Gastrointestinal disorders) | 0 (0) | 1 (1) | 0 (0)
Mouth swelling (Gastrointestinal disorders) | 0 (0) | 1 (1) | 0 (0)
Nausea (Gastrointestinal disorders) | 15 (15) | 4 (4) | 0 (0)
Stomatitis (Gastrointestinal disorders) | 0 (0) | 0 (0) | 1 (1)
Toothache (Gastrointestinal disorders) | 1 (1) | 1 (1) | 0 (0)
Vomiting (Gastrointestinal disorders) | 7 (8) | 3 (3) | 0 (0)
Adverse drug reaction (General disorders) | 1 (1) | 0 (0) | 0 (0)
Asthenia (General disorders) | 4 (4) | 2 (2) | 1 (1)
Chest discomfort (General disorders) | 1 (1) | 0 (0) | 0 (0)
Chest pain (General disorders) | 1 (1) | 1 (1) | 0 (0)
Chills (General disorders) | 1 (1) | 0 (0) | 1 (1)
Early satiety (General disorders) | 0 (0) | 1 (1) | 0 (0)
Face oedema (General disorders) | 0 (0) | 1 (1) | 0 (0)
Fatigue (General disorders) | 5 (6) | 5 (5) | 1 (1)
Feeling abnormal (General disorders) | 0 (0) | 1 (1) | 0 (0)
Gait disturbance (General disorders) | 1 (1) | 0 (0) | 0 (0)
General physical health deterioration (General disorders) | 1 (1) | 0 (0) | 0 (0)
Hyperthermia (General disorders) | 0 (0) | 1 (1) | 0 (0)
Influenza like illness (General disorders) | 0 (0) | 1 (1) | 0 (0)
Infusion site pain (General disorders) | 0 (0) | 0 (0) | 1 (1)
Infusion site swelling (General disorders) | 0 (0) | 1 (2) | 0 (0)
Injection site pain (General disorders) | 0 (0) | 1 (1) | 0 (0)
Injection site pruritus (General disorders) | 1 (1) | 0 (0) | 0 (0)
Malaise (General disorders) | 0 (0) | 1 (1) | 0 (0)
Medical device site reaction (General disorders) | 1 (1) | 0 (0) | 0 (0)
Oedema peripheral (General disorders) | 0 (0) | 3 (3) | 0 (0)
Peripheral swelling (General disorders) | 1 (1) | 0 (0) | 0 (0)
Precancerous condition (General disorders) | 0 (0) | 1 (2) | 0 (0)
Pyrexia (General disorders) | 1 (1) | 2 (2) | 0 (0)
Soft tissue inflammation (General disorders) | 1 (1) | 0 (0) | 0 (0)
Systemic inflammatory response syndrome (General disorders) | 0 (0) | 1 (1) | 0 (0)
Vessel puncture site bruise (General disorders) | 0 (0) | 2 (3) | 0 (0)
Bile duct stone (Hepatobiliary disorders) | 0 (0) | 1 (1) | 0 (0)
Cholecystitis (Hepatobiliary disorders) | 0 (0) | 1 (1) | 0 (0)
Cholelithiasis (Hepatobiliary disorders) | 1 (1) | 0 (0) | 0 (0)
Drug hypersensitivity (Immune system disorders) | 0 (0) | 0 (0) | 1 (1)
Hypersensitivity (Immune system disorders) | 0 (0) | 1 (1) | 0 (0)
Seasonal allergy (Immune system disorders) | 1 (1) | 0 (0) | 1 (1)
Acute sinusitis (Infections and infestations) | 0 (0) | 0 (0) | 1 (1)
Asymptomatic covid-19 (Infections and infestations) | 0 (0) | 1 (1) | 0 (0)
Bronchitis (Infections and infestations) | 4 (4) | 2 (2) | 0 (0)
Bronchitis viral (Infections and infestations) | 1 (1) | 0 (0) | 0 (0)
Cellulitis (Infections and infestations) | 2 (2) | 2 (2) | 2 (2)
Clostridium difficile colitis (Infections and infestations) | 1 (1) | 1 (1) | 0 (0)
Conjunctivitis (Infections and infestations) | 0 (0) | 2 (2) | 0 (0)
Covid-19 (Infections and infestations) | 2 (2) | 1 (1) | 0 (0)
Eyelid infection (Infections and infestations) | 0 (0) | 1 (1) | 0 (0)
Fungal infection (Infections and infestations) | 1 (1) | 0 (0) | 0 (0)
Fungal skin infection (Infections and infestations) | 0 (0) | 2 (2) | 0 (0)
Gastroenteritis (Infections and infestations) | 0 (0) | 2 (2) | 0 (0)
Gastrointestinal viral infection (Infections and infestations) | 0 (0) | 1 (1) | 0 (0)
Gingivitis (Infections and infestations) | 0 (0) | 1 (1) | 0 (0)
Herpes zoster (Infections and infestations) | 0 (0) | 3 (3) | 1 (1)
Hordeolum (Infections and infestations) | 1 (1) | 0 (0) | 0 (0)
Influenza (Infections and infestations) | 2 (2) | 1 (1) | 0 (0)
Labyrinthitis (Infections and infestations) | 0 (0) | 0 (0) | 1 (1)
Laryngitis (Infections and infestations) | 1 (1) | 1 (1) | 0 (0)
Localised infection (Infections and infestations) | 0 (0) | 1 (1) | 0 (0)
Lower respiratory tract infection (Infections and infestations) | 1 (1) | 0 (0) | 0 (0)
Lyme disease (Infections and infestations) | 1 (1) | 2 (2) | 0 (0)
Nasopharyngitis (Infections and infestations) | 6 (7) | 6 (7) | 0 (0)
Onychomycosis (Infections and infestations) | 0 (0) | 1 (1) | 0 (0)
Oral herpes (Infections and infestations) | 1 (1) | 0 (0) | 0 (0)
Otitis media acute (Infections and infestations) | 0 (0) | 0 (0) | 1 (1)
Pneumonia (Infections and infestations) | 3 (3) | 4 (4) | 1 (1)
Postoperative wound infection (Infections and infestations) | 0 (0) | 0 (0) | 1 (1)
Root canal infection (Infections and infestations) | 0 (0) | 0 (0) | 1 (1)
Sinusitis (Infections and infestations) | 1 (1) | 2 (2) | 0 (0)
Skin candida (Infections and infestations) | 0 (0) | 0 (0) | 1 (1)
Skin infection (Infections and infestations) | 2 (2) | 0 (0) | 0 (0)
Testicular abscess (Infections and infestations) | 0/63 (0) | 1/61 (1) | 0/3 (0)
Tooth abscess (Infections and infestations) | 1 (1) | 1 (1) | 0 (0)
Tooth infection (Infections and infestations) | 0 (0) | 1 (1) | 0 (0)
Upper respiratory tract infection (Infections and infestations) | 9 (11) | 9 (10) | 2 (2)
Urinary tract infection (Infections and infestations) | 13 (22) | 4 (5) | 2 (2)
Viral upper respiratory tract infection (Infections and infestations) | 1 (1) | 1 (1) | 0 (0)
Animal bite (Injury, poisoning and procedural complications) | 0 (0) | 2 (2) | 0 (0)
Arthropod bite (Injury, poisoning and procedural complications) | 1 (1) | 2 (2) | 0 (0)
Arthropod sting (Injury, poisoning and procedural complications) | 2 (3) | 1 (1) | 0 (0)
Bone contusion (Injury, poisoning and procedural complications) | 2 (2) | 1 (1) | 0 (0)
Buttock injury (Injury, poisoning and procedural complications) | 0 (0) | 1 (1) | 0 (0)
Cataract operation complication (Injury, poisoning and procedural complications) | 1 (1) | 0 (0) | 0 (0)
Clavicle fracture (Injury, poisoning and procedural complications) | 1 (1) | 0 (0) | 0 (0)
Contusion (Injury, poisoning and procedural complications) | 0 (0) | 11 (12) | 0 (0)
Eye contusion (Injury, poisoning and procedural complications) | 0 (0) | 1 (1) | 0 (0)
Facial bones fracture (Injury, poisoning and procedural complications) | 1 (1) | 1 (1) | 0 (0)
Fall (Injury, poisoning and procedural complications) | 19 (23) | 21 (30) | 1 (1)
Foot fracture (Injury, poisoning and procedural complications) | 1 (1) | 0 (0) | 0 (0)
Hand fracture (Injury, poisoning and procedural complications) | 0 (0) | 1 (1) | 0 (0)
Head injury (Injury, poisoning and procedural complications) | 1 (1) | 2 (2) | 0 (0)
Infusion related reaction (Injury, poisoning and procedural complications) | 8 (29) | 0 (0) | 1 (3)
Joint injury (Injury, poisoning and procedural complications) | 0 (0) | 1 (1) | 0 (0)
Ligament sprain (Injury, poisoning and procedural complications) | 1 (1) | 4 (5) | 1 (1)
Limb injury (Injury, poisoning and procedural complications) | 1 (1) | 0 (0) | 0 (0)
Lumbar vertebral fracture (Injury, poisoning and procedural complications) | 0 (0) | 1 (1) | 0 (0)
Meniscus injury (Injury, poisoning and procedural complications) | 1 (1) | 1 (1) | 1 (1)
Muscle strain (Injury, poisoning and procedural complications) | 0 (0) | 2 (2) | 0 (0)
Procedural pain (Injury, poisoning and procedural complications) | 0 (0) | 1 (1) | 0 (0)
Radiation injury (Injury, poisoning and procedural complications) | 0 (0) | 1 (1) | 0 (0)
Radius fracture (Injury, poisoning and procedural complications) | 0 (0) | 1 (1) | 0 (0)
Rib fracture (Injury, poisoning and procedural complications) | 1 (1) | 1 (1) | 0 (0)
Road traffic accident (Injury, poisoning and procedural complications) | 0 (0) | 2 (2) | 0 (0)
Skin abrasion (Injury, poisoning and procedural complications) | 4 (4) | 3 (4) | 1 (1)
Skin injury (Injury, poisoning and procedural complications) | 1 (1) | 0 (0) | 0 (0)
Skin laceration (Injury, poisoning and procedural complications) | 2 (2) | 4 (4) | 0 (0)
Spinal compression fracture (Injury, poisoning and procedural complications) | 0 (0) | 1 (1) | 0 (0)
Synovial rupture (Injury, poisoning and procedural complications) | 1 (1) | 0 (0) | 0 (0)
Tendon rupture (Injury, poisoning and procedural complications) | 1 (1) | 0 (0) | 0 (0)
Tooth fracture (Injury, poisoning and procedural complications) | 1 (1) | 0 (0) | 0 (0)
Traumatic haematoma (Injury, poisoning and procedural complications) | 1 (1) | 1 (1) | 0 (0)
Vaccination complication (Injury, poisoning and procedural complications) | 1 (1) | 0 (0) | 0 (0)
Wound (Injury, poisoning and procedural complications) | 2 (2) | 1 (2) | 0 (0)
Wrist fracture (Injury, poisoning and procedural complications) | 2 (2) | 0 (0) | 0 (0)
Alanine aminotransferase increased (Investigations) | 0 (0) | 1 (1) | 0 (0)
Aspartate aminotransferase increased (Investigations) | 0 (0) | 2 (2) | 0 (0)
Bacterial test positive (Investigations) | 1 (1) | 0 (0) | 0 (0)
Biopsy skin (Investigations) | 1 (1) | 0 (0) | 0 (0)
Blood alkaline phosphatase increased (Investigations) | 0 (0) | 1 (2) | 0 (0)
Blood creatine phosphokinase increased (Investigations) | 0 (0) | 0 (0) | 1 (1)
Blood glucose increased (Investigations) | 0 (0) | 1 (1) | 0 (0)
Blood potassium decreased (Investigations) | 0 (0) | 1 (1) | 0 (0)
Blood pressure increased (Investigations) | 1 (1) | 1 (1) | 0 (0)
Blood pressure systolic increased (Investigations) | 1 (1) | 1 (1) | 0 (0)
C-reactive protein increased (Investigations) | 1 (1) | 0 (0) | 0 (0)
Cardiac murmur (Investigations) | 1 (1) | 1 (1) | 0 (0)
Creatinine renal clearance decreased (Investigations) | 1 (1) | 0 (0) | 0 (0)
Electrocardiogram pr shortened (Investigations) | 0 (0) | 0 (0) | 1 (1)
Electrocardiogram qt prolonged (Investigations) | 2 (3) | 0 (0) | 0 (0)
Haemoglobin decreased (Investigations) | 1 (1) | 0 (0) | 0 (0)
Heart rate irregular (Investigations) | 1 (1) | 1 (1) | 0 (0)
Liver function test increased (Investigations) | 0 (0) | 0 (0) | 1 (1)
Lymphocyte morphology abnormal (Investigations) | 1 (1) | 0 (0) | 0 (0)
Occult blood positive (Investigations) | 1 (1) | 0 (0) | 0 (0)
Platelet count decreased (Investigations) | 0 (0) | 1 (1) | 0 (0)
Prostatic specific antigen increased (Investigations) | 1/63 (1) | 0/61 (0) | 0/3 (0)
Qrs axis abnormal (Investigations) | 1 (1) | 1 (1) | 0 (0)
Urine leukocyte esterase positive (Investigations) | 0 (0) | 0 (0) | 1 (1)
Weight decreased (Investigations) | 4 (4) | 4 (4) | 0 (0)
Weight increased (Investigations) | 1 (1) | 0 (0) | 0 (0)
Decreased appetite (Metabolism and nutrition disorders) | 2 (2) | 2 (2) | 0 (0)
Dehydration (Metabolism and nutrition disorders) | 2 (2) | 4 (4) | 0 (0)
Glucose tolerance impaired (Metabolism and nutrition disorders) | 1 (1) | 0 (0) | 0 (0)
Gout (Metabolism and nutrition disorders) | 0 (0) | 2 (2) | 0 (0)
Hypercholesterolaemia (Metabolism and nutrition disorders) | 1 (1) | 1 (1) | 0 (0)
Hyperglycaemia (Metabolism and nutrition disorders) | 1 (1) | 0 (0) | 0 (0)
Hyperkalaemia (Metabolism and nutrition disorders) | 1 (1) | 0 (0) | 0 (0)
Hyperuricaemia (Metabolism and nutrition disorders) | 0 (0) | 2 (2) | 0 (0)
Hypocalcaemia (Metabolism and nutrition disorders) | 1 (1) | 1 (1) | 0 (0)
Hypoglycaemia (Metabolism and nutrition disorders) | 2 (2) | 0 (0) | 0 (0)
Hypokalaemia (Metabolism and nutrition disorders) | 0 (0) | 5 (6) | 0 (0)
Hypomagnesaemia (Metabolism and nutrition disorders) | 1 (1) | 0 (0) | 0 (0)
Hyponatraemia (Metabolism and nutrition disorders) | 2 (2) | 2 (2) | 0 (0)
Lactic acidosis (Metabolism and nutrition disorders) | 1 (1) | 0 (0) | 0 (0)
Malnutrition (Metabolism and nutrition disorders) | 1 (1) | 0 (0) | 0 (0)
Overweight (Metabolism and nutrition disorders) | 1 (1) | 0 (0) | 0 (0)
Type 2 diabetes mellitus (Metabolism and nutrition disorders) | 0 (0) | 2 (2) | 0 (0)
Vitamin b12 deficiency (Metabolism and nutrition disorders) | 1 (1) | 0 (0) | 0 (0)
Arthralgia (Musculoskeletal and connective tissue disorders) | 12 (14) | 10 (10) | 3 (3)
Arthritis (Musculoskeletal and connective tissue disorders) | 2 (3) | 2 (2) | 0 (0)
Back pain (Musculoskeletal and connective tissue disorders) | 4 (6) | 4 (4) | 1 (1)
Bursitis (Musculoskeletal and connective tissue disorders) | 2 (2) | 3 (4) | 0 (0)
Coccydynia (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1) | 0 (0)
Facet joint syndrome (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0) | 0 (0)
Intervertebral disc protrusion (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 1 (1)
Jaw disorder (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0) | 0 (0)
Joint effusion (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0) | 0 (0)
Joint stiffness (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1) | 0 (0)
Joint swelling (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 1 (1)
Mucoid degeneration of the anterior cruciate ligament (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0) | 0 (0)
Muscle atrophy (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1) | 0 (0)
Muscle spasms (Musculoskeletal and connective tissue disorders) | 1 (1) | 2 (3) | 0 (0)
Muscle twitching (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1) | 0 (0)
Muscular weakness (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1) | 0 (0)
Musculoskeletal chest pain (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0) | 0 (0)
Musculoskeletal pain (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1) | 0 (0)
Neck pain (Musculoskeletal and connective tissue disorders) | 1 (1) | 3 (3) | 0 (0)
Osteoarthritis (Musculoskeletal and connective tissue disorders) | 2 (2) | 1 (1) | 0 (0)
Osteochondritis (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0) | 0 (0)
Pain in extremity (Musculoskeletal and connective tissue disorders) | 5 (5) | 3 (3) | 1 (1)
Plantar fasciitis (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 1 (1)
Rheumatoid arthritis (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0) | 0 (0)
Rotator cuff syndrome (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1) | 0 (0)
Sacroiliitis (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1) | 0 (0)
Spinal osteoarthritis (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1) | 0 (0)
Spinal stenosis (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0) | 0 (0)
Synovial cyst (Musculoskeletal and connective tissue disorders) | 1 (2) | 1 (1) | 0 (0)
Temporomandibular joint syndrome (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0) | 0 (0)
Tendonitis (Musculoskeletal and connective tissue disorders) | 1 (1) | 1 (1) | 0 (0)
Trigger finger (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1) | 0 (0)
Atypical fibroxanthoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0) | 0 (0)
Basal cell carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 3 (3) | 4 (4) | 0 (0)
Benign lung neoplasm (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 2 (2) | 0 (0) | 0 (0)
Bowen's disease (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 1 (1) | 0 (0)
Dysplastic naevus (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (2) | 0 (0) | 0 (0)
Enchondromatosis (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 0 (0) | 1 (1)
Keratoacanthoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 1 (1) | 0 (0)
Lip neoplasm (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 1 (1) | 0 (0)
Lung adenocarcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0) | 0 (0)
Malignant melanoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 1 (1) | 0 (0)
Neuroma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0) | 0 (0)
Non-hodgkin's lymphoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 1 (1) | 0 (0)
Prostate cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0/63 (0) | 1/61 (1) | 0/3 (0)
Seborrhoeic keratosis (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0) | 0 (0)
Skin papilloma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 1 (1) | 0 (0)
Squamous cell carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 3 (3) | 1 (1) | 0 (0)
Squamous cell carcinoma of skin (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 2 (2) | 0 (0)
Ageusia (Nervous system disorders) | 0 (0) | 1 (1) | 0 (0)
Amyloid related imaging abnormality-microhaemorrhages and haemosiderin deposits (Nervous system disorders) | 11 (14) | 4 (5) | 1 (1)
Amyloid related imaging abnormality-oedema/effusion (Nervous system disorders) | 33 (43) | 1 (2) | 4 (4)
Balance disorder (Nervous system disorders) | 1 (1) | 3 (4) | 1 (1)
Burning sensation (Nervous system disorders) | 0 (0) | 1 (1) | 0 (0)
Cerebellar microhaemorrhage (Nervous system disorders) | 2 (3) | 0 (0) | 0 (0)
Cerebral infarction (Nervous system disorders) | 1 (1) | 0 (0) | 0 (0)
Cerebral microhaemorrhage (Nervous system disorders) | 10 (18) | 3 (6) | 2 (2)
Cerebrovascular accident (Nervous system disorders) | 0 (0) | 0 (0) | 1 (1)
Cluster headache (Nervous system disorders) | 0 (0) | 1 (1) | 0 (0)
Cognitive disorder (Nervous system disorders) | 1 (1) | 1 (1) | 0 (0)
Dementia alzheimer's type (Nervous system disorders) | 1 (1) | 1 (1) | 0 (0)
Dizziness (Nervous system disorders) | 11 (16) | 14 (16) | 4 (4)
Dizziness postural (Nervous system disorders) | 0 (0) | 1 (1) | 0 (0)
Drug withdrawal headache (Nervous system disorders) | 1 (1) | 0 (0) | 0 (0)
Dysarthria (Nervous system disorders) | 0 (0) | 0 (0) | 1 (1)
Encephalopathy (Nervous system disorders) | 0 (0) | 1 (1) | 0 (0)
Essential tremor (Nervous system disorders) | 2 (2) | 0 (0) | 0 (0)
Gliosis (Nervous system disorders) | 1 (1) | 0 (0) | 0 (0)
Head discomfort (Nervous system disorders) | 1 (1) | 0 (0) | 0 (0)
Headache (Nervous system disorders) | 10 (11) | 15 (17) | 0 (0)
Hemiparesis (Nervous system disorders) | 0 (0) | 0 (0) | 1 (1)
Hypoaesthesia (Nervous system disorders) | 0 (0) | 2 (2) | 1 (1)
Intraventricular haemorrhage (Nervous system disorders) | 0 (0) | 1 (1) | 0 (0)
Lacunar infarction (Nervous system disorders) | 0 (0) | 2 (3) | 0 (0)
Lethargy (Nervous system disorders) | 1 (1) | 0 (0) | 0 (0)
Loss of consciousness (Nervous system disorders) | 0 (0) | 1 (1) | 0 (0)
Memory impairment (Nervous system disorders) | 0 (0) | 1 (1) | 0 (0)
Migraine (Nervous system disorders) | 1 (1) | 0 (0) | 0 (0)
Neuralgia (Nervous system disorders) | 1 (1) | 0 (0) | 1 (1)
Occipital neuralgia (Nervous system disorders) | 1 (1) | 0 (0) | 0 (0)
Paraesthesia (Nervous system disorders) | 1 (1) | 0 (0) | 2 (2)
Parkinson's disease (Nervous system disorders) | 0 (0) | 1 (1) | 0 (0)
Patient elopement (Nervous system disorders) | 1 (1) | 0 (0) | 0 (0)
Peripheral sensorimotor neuropathy (Nervous system disorders) | 1 (1) | 1 (1) | 0 (0)
Polyneuropathy (Nervous system disorders) | 1 (1) | 0 (0) | 0 (0)
Presyncope (Nervous system disorders) | 3 (4) | 0 (0) | 0 (0)
Resting tremor (Nervous system disorders) | 0 (0) | 1 (1) | 0 (0)
Sciatica (Nervous system disorders) | 1 (1) | 1 (1) | 1 (1)
Sensory loss (Nervous system disorders) | 1 (1) | 0 (0) | 0 (0)
Superficial siderosis of central nervous system (Nervous system disorders) | 18 (23) | 4 (4) | 3 (4)
Syncope (Nervous system disorders) | 3 (4) | 5 (6) | 0 (0)
Transient ischaemic attack (Nervous system disorders) | 0 (0) | 1 (1) | 0 (0)
Tremor (Nervous system disorders) | 1 (1) | 1 (1) | 1 (1)
Trigeminal neuralgia (Nervous system disorders) | 0 (0) | 0 (0) | 1 (1)
Abnormal dreams (Psychiatric disorders) | 0 (0) | 1 (1) | 0 (0)
Adjustment disorder (Psychiatric disorders) | 0 (0) | 0 (0) | 1 (1)
Agitation (Psychiatric disorders) | 0 (0) | 5 (5) | 1 (1)
Anxiety (Psychiatric disorders) | 7 (8) | 3 (3) | 1 (1)
Confusional state (Psychiatric disorders) | 3 (3) | 2 (2) | 0 (0)
Delusion (Psychiatric disorders) | 2 (2) | 2 (3) | 1 (1)
Depressed mood (Psychiatric disorders) | 0 (0) | 3 (3) | 0 (0)
Depression (Psychiatric disorders) | 6 (6) | 9 (9) | 1 (1)
Disinhibition (Psychiatric disorders) | 0 (0) | 1 (1) | 0 (0)
Emotional disorder (Psychiatric disorders) | 0 (0) | 1 (1) | 0 (0)
Hallucination (Psychiatric disorders) | 1 (1) | 1 (1) | 1 (1)
Initial insomnia (Psychiatric disorders) | 1 (1) | 0 (0) | 0 (0)
Insomnia (Psychiatric disorders) | 1 (1) | 3 (3) | 0 (0)
Irritability (Psychiatric disorders) | 1 (1) | 2 (2) | 0 (0)
Nightmare (Psychiatric disorders) | 2 (2) | 2 (2) | 0 (0)
Procedural anxiety (Psychiatric disorders) | 0 (0) | 1 (1) | 0 (0)
Rapid eye movements sleep abnormal (Psychiatric disorders) | 0 (0) | 2 (2) | 0 (0)
Suicidal ideation (Psychiatric disorders) | 0 (0) | 4 (6) | 0 (0)
Acute kidney injury (Renal and urinary disorders) | 2 (2) | 2 (2) | 0 (0)
Dysuria (Renal and urinary disorders) | 0 (0) | 1 (1) | 0 (0)
Glycosuria (Renal and urinary disorders) | 1 (1) | 0 (0) | 0 (0)
Haematuria (Renal and urinary disorders) | 0 (0) | 1 (1) | 0 (0)
Hydronephrosis (Renal and urinary disorders) | 1 (1) | 0 (0) | 0 (0)
Hypertonic bladder (Renal and urinary disorders) | 0 (0) | 2 (2) | 0 (0)
Nephrolithiasis (Renal and urinary disorders) | 1 (1) | 0 (0) | 0 (0)
Pollakiuria (Renal and urinary disorders) | 2 (2) | 0 (0) | 0 (0)
Renal cyst (Renal and urinary disorders) | 1 (1) | 0 (0) | 0 (0)
Renal failure (Renal and urinary disorders) | 0 (0) | 1 (1) | 0 (0)
Urge incontinence (Renal and urinary disorders) | 0 (0) | 0 (0) | 1 (1)
Urinary incontinence (Renal and urinary disorders) | 3 (3) | 3 (3) | 0 (0)
Urinary retention (Renal and urinary disorders) | 1 (1) | 0 (0) | 0 (0)
Urinary tract obstruction (Renal and urinary disorders) | 0 (0) | 1 (1) | 0 (0)
Benign prostatic hyperplasia (Reproductive system and breast disorders) | 1/63 (1) | 1/61 (1) | 0/3 (0)
Uterine disorder (Reproductive system and breast disorders) | 1/68 (1) | 0/64 (0) | 0/12 (0)
Atelectasis (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 1 (1) | 0 (0)
Cough (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1) | 0 (0)
Dysphonia (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1) | 0 (0)
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 3 (4) | 0 (0)
Dyspnoea exertional (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 2 (2) | 0 (0)
Haemoptysis (Respiratory, thoracic and mediastinal disorders) | 2 (2) | 0 (0) | 0 (0)
Hiccups (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0) | 0 (0)
Hypoxia (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0) | 0 (0)
Oropharyngeal pain (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 1 (1) | 0 (0)
Pharyngeal swelling (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1) | 0 (0)
Pleural effusion (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1) | 0 (0)
Productive cough (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 1 (1)
Pulmonary mass (Respiratory, thoracic and mediastinal disorders) | 2 (2) | 0 (0) | 1 (1)
Rhinitis allergic (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1) | 0 (0)
Rhinorrhoea (Respiratory, thoracic and mediastinal disorders) | 2 (2) | 0 (0) | 0 (0)
Sinus congestion (Respiratory, thoracic and mediastinal disorders) | 2 (2) | 0 (0) | 1 (1)
Sleep apnoea syndrome (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 1 (1) | 0 (0)
Upper-airway cough syndrome (Respiratory, thoracic and mediastinal disorders) | 2 (2) | 0 (0) | 0 (0)
Actinic keratosis (Skin and subcutaneous tissue disorders) | 1 (3) | 0 (0) | 1 (1)
Alopecia (Skin and subcutaneous tissue disorders) | 2 (2) | 0 (0) | 0 (0)
Angioedema (Skin and subcutaneous tissue disorders) | 0 (0) | 1 (1) | 1 (1)
Dermatitis (Skin and subcutaneous tissue disorders) | 1 (1) | 1 (1) | 0 (0)
Dermatitis allergic (Skin and subcutaneous tissue disorders) | 1 (1) | 0 (0) | 0 (0)
Dermatitis bullous (Skin and subcutaneous tissue disorders) | 1 (5) | 0 (0) | 0 (0)
Dermatitis contact (Skin and subcutaneous tissue disorders) | 1 (1) | 1 (1) | 0 (0)
Ecchymosis (Skin and subcutaneous tissue disorders) | 0 (0) | 1 (1) | 0 (0)
Eczema (Skin and subcutaneous tissue disorders) | 0 (0) | 1 (1) | 1 (1)
Erythema (Skin and subcutaneous tissue disorders) | 1 (1) | 0 (0) | 0 (0)
Ingrowing nail (Skin and subcutaneous tissue disorders) | 1 (1) | 0 (0) | 0 (0)
Lentigo (Skin and subcutaneous tissue disorders) | 0 (0) | 1 (1) | 0 (0)
Petechiae (Skin and subcutaneous tissue disorders) | 0 (0) | 1 (1) | 0 (0)
Precancerous skin lesion (Skin and subcutaneous tissue disorders) | 0 (0) | 1 (3) | 0 (0)
Pruritus (Skin and subcutaneous tissue disorders) | 1 (1) | 0 (0) | 0 (0)
Purpura (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 1 (1)
Rash (Skin and subcutaneous tissue disorders) | 0 (0) | 6 (8) | 2 (2)
Rash macular (Skin and subcutaneous tissue disorders) | 0 (0) | 1 (1) | 0 (0)
Seborrhoeic dermatitis (Skin and subcutaneous tissue disorders) | 1 (1) | 1 (1) | 0 (0)
Skin discolouration (Skin and subcutaneous tissue disorders) | 0 (0) | 1 (1) | 0 (0)
Skin hyperpigmentation (Skin and subcutaneous tissue disorders) | 1 (2) | 0 (0) | 0 (0)
Skin hypopigmentation (Skin and subcutaneous tissue disorders) | 0 (0) | 1 (1) | 0 (0)
Skin lesion (Skin and subcutaneous tissue disorders) | 0 (0) | 3 (3) | 0 (0)
Skin ulcer (Skin and subcutaneous tissue disorders) | 0 (0) | 1 (1) | 0 (0)
Transient acantholytic dermatosis (Skin and subcutaneous tissue disorders) | 1 (1) | 0 (0) | 0 (0)
Urticaria (Skin and subcutaneous tissue disorders) | 1 (1) | 0 (0) | 0 (0)
Blepharorrhaphy (Surgical and medical procedures) | 1 (1) | 0 (0) | 0 (0)
Cancer surgery (Surgical and medical procedures) | 0 (0) | 1 (1) | 0 (0)
Cardiac pacemaker insertion (Surgical and medical procedures) | 1 (1) | 0 (0) | 0 (0)
Cardiac pacemaker replacement (Surgical and medical procedures) | 1 (1) | 1 (1) | 0 (0)
Cataract operation (Surgical and medical procedures) | 3 (4) | 2 (3) | 1 (2)
Cryotherapy (Surgical and medical procedures) | 1 (1) | 0 (0) | 0 (0)
Dental implantation (Surgical and medical procedures) | 1 (1) | 0 (0) | 0 (0)
Endodontic procedure (Surgical and medical procedures) | 0 (0) | 1 (1) | 0 (0)
Intraocular lens implant (Surgical and medical procedures) | 1 (1) | 0 (0) | 0 (0)
Lens extraction (Surgical and medical procedures) | 1 (1) | 0 (0) | 0 (0)
Medical device removal (Surgical and medical procedures) | 0 (0) | 0 (0) | 1 (1)
Precancerous lesion excision (Surgical and medical procedures) | 0 (0) | 1 (1) | 0 (0)
Shoulder arthroplasty (Surgical and medical procedures) | 0 (0) | 1 (1) | 1 (1)
Skin cryotherapy (Surgical and medical procedures) | 1 (1) | 1 (1) | 0 (0)
Skin neoplasm excision (Surgical and medical procedures) | 0 (0) | 0 (0) | 1 (1)
Spinal operation (Surgical and medical procedures) | 0 (0) | 0 (0) | 1 (1)
Tooth extraction (Surgical and medical procedures) | 1 (1) | 6 (6) | 0 (0)
Vertebroplasty (Surgical and medical procedures) | 0 (0) | 1 (1) | 0 (0)
Vitrectomy (Surgical and medical procedures) | 0 (0) | 1 (1) | 0 (0)
Hot flush (Vascular disorders) | 3 (3) | 0 (0) | 0 (0)
Hypertension (Vascular disorders) | 3 (3) | 6 (6) | 0 (0)
Hypertensive urgency (Vascular disorders) | 0 (0) | 1 (1) | 0 (0)
Hypotension (Vascular disorders) | 4 (4) | 2 (2) | 0 (0)
Labile hypertension (Vascular disorders) | 0 (0) | 0 (0) | 1 (1)
Orthostatic hypotension (Vascular disorders) | 2 (2) | 0 (0) | 0 (0)
Peripheral venous disease (Vascular disorders) | 1 (1) | 0 (0) | 0 (0)
Poor venous access (Vascular disorders) | 3 (3) | 1 (1) | 0 (0)

LIMITATIONS AND CAVEATS:
As per protocol amendment (d) approved on Oct 9, 2018, donanemab in combination with LY3202626 (donanemab-C) arm discontinued as there was a low probability of identifying a statistically significant effect of 12mg of LY3202626 slowing cognitive decline. Clinical efficacy was not reported for this group.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
The only disclosure restriction on the PI is that the sponsor can review results communications prior to public release and can embargo communications regarding trial results for a period that is more than 30 days but less than or equal to 90 days from the time submitted to the sponsor for review. The sponsor cannot require changes to the communication and cannot extend the embargo.

DOCUMENTS (2):
  • Study Protocol (2018-10-09): https://cdn.clinicaltrials.gov/large-docs/03/NCT03367403/Prot_000.pdf
  • Statistical Analysis Plan (2020-12-07): https://cdn.clinicaltrials.gov/large-docs/03/NCT03367403/SAP_001.pdf